CLINICAL TRIAL: NCT02549027
Title: A Crossover Study to Evaluate the Effects of Single Doses of MK-1064 and MK-6096 on Polysomnography (PSG)
Brief Title: A Study to Evaluate the Effects of Single Doses of MK-1064 and MK-6096 on Polysomnography (PSG) (MK-1064-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1064-003
Record Dates: First submitted 2015-09-11; First posted 2015-09-14 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Polysomnography
MeSH Terms: interventions — MK-6096

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence (MK-1064): 50 mg→250 mg→Placebo→120 mg (Experimental): For overall study population, 5 participants each were to be allocated to one of 4 sequences. In this sequence, participants received the following: Period 1 - single dose of 50 mg MK-1064, Period 2 - single dose of 250 mg MK-1064, Period 3 - single dose of placebo, Period 4 - single dose of 120 mg MK-1064. Participants completing the first 4 periods also were to receive the following: Period 5 - single dose of 20 mg MK-6096 or placebo, in an 18:2 ratio for overall study population, according to separate allocation. There was a minimum 7-day washout between doses.
  Interventions: Drug: MK-1064; Drug: MK-6096; Drug: Placebo
- Sequence (MK-1064): Placebo→50 mg→120 mg→250 mg (Experimental): For overall study population, 5 participants each were to be allocated to one of 4 sequences. In this sequence, participants received the following: Period 1 - single dose of placebo, Period 2 - single dose of 50 mg MK-1064, Period 3 - single dose of 120 mg MK-1064, Period 4 - single dose of 250 mg MK-1064. Participants completing the first 4 periods also were to receive the following: Period 5 - single dose of 20 mg MK-6096 or placebo, in an 18:2 ratio for overall study population, according to separate allocation. There was a minimum 7-day washout between doses.
  Interventions: Drug: MK-1064; Drug: MK-6096; Drug: Placebo
- Sequence (MK-1064): 120 mg→Placebo→250 mg→50 mg (Experimental): For overall study population, 5 participants each were to be allocated to one of 4 sequences. In this sequence, participants received the following: Period 1 - single dose of 120 mg MK-1064, Period 2 - single dose of placebo, Period 3 - single dose of 250 mg MK-1064, Period 4 - single dose of 50 mg MK-1064. Participants completing the first 4 periods also were to receive the following: Period 5 - single dose of 20 mg MK-6096 or placebo, in an 18:2 ratio for overall study population, according to separate allocation. There was a minimum 7-day washout between doses.
  Interventions: Drug: MK-1064; Drug: MK-6096; Drug: Placebo
- Sequence (MK-1064): 250 mg→120 mg→50 mg→Placebo (Experimental): For overall study population, 5 participants each were to be allocated to one of 4 sequences. In this sequence, participants received the following: Period 1 - single dose of 250 mg MK-1064, Period 2 - single dose of 120 mg MK-1064, Period 3 - single dose of 50 mg MK-1064, Period 4 - single dose of placebo. Participants completing the first 4 periods also were to receive the following: Period 5 - single dose of 20 mg MK-6096 or placebo, in an 18:2 ratio for overall study population, according to separate allocation. There was a minimum 7-day washout between doses.
  Interventions: Drug: MK-1064; Drug: MK-6096; Drug: Placebo

INTERVENTIONS:
Drug: MK-1064 — Oral MK-1064 tablets (10 and 50 mg strengths)
Drug: MK-6096 — Oral MK-6096 tablets (5 mg strength)
Drug: Placebo — Oral placebo tablets (matching active MK-1064 tablets, matching active MK-6096 tablets)

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled, 5-period crossover study is to assess the effect of single oral doses of MK-1064 on latency to persistent sleep (LPS) as measured by polysomnography (PSG) in healthy young male participants, and to evaluate the safety and tolerability of single oral doses of MK-1064 and MK-6096 in healthy young male participants. The primary efficacy hypothesis is that at least one dose of MK-1064 is superior to placebo in decreasing LPS in healthy male participants as assessed by PSG.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≤31 kg/m^2
* In good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests
* Nonsmoker and has not used nicotine or nicotine-containing products for at least 6 months
* No history of any sleep disorder
* Has not used prescription or over the counter sedation or alerting medication in 4 weeks prior to screening
* Participant has a usual bedtime between 8:00 PM and 12:00 AM
* Participant has total sleep duration of ≥6.5 and ≤9 hours during the 4 weeks prior to screening
* Male participants with female partner(s) of child-bearing potential must agree to use a medically acceptable method of contraception during the study and for 90 days after the last dose of study drug

Exclusion Criteria:

* Mentally or legally incapacitated, significant emotional problems at screening or expected during the conduct of the study or history of a clinically significant psychiatric disorder within the last 10 years
* History of any persistent sleep abnormality (including difficulty falling asleep, difficulty staying asleep) lasting for 3 months or more, or history of obstructive sleep apnea, restless leg syndrome, or narcolepsy
* History of clinically significant sleep disorders within the last 5 years
* History of circadian rhythm sleep disorder, clinically important parasomnia, or primary insomnia
* History of repeated falls or fractures secondary to falling within the past 2 years
* Participant works a night shift and is not able to avoid night shift work a minimum of 1 week prior to screening and for the duration of the study
* Participant has traveled across 3 or more time zones (transmeridian travel) in the last 2 weeks prior to study
* Is a regular user of sedative-hypnotic agents
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of stroke, peripheral neuropathy, chronic seizures or other clinically significant neurological disorder or cognitive impairment
* History of cancer
* History of cataplexy
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies, beginning approximately 2 weeks prior to administration of the initial dose of study drug and throughout the study
* Participant consumes >3 servings of alcohol a day
* Participant consumes >6 caffeine servings a day
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to screening, or participated in another investigational study within 3 months prior to first dose of study drug
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is currently a regular user of any illicit drugs or has a history of drug (including alcohol) abuse within 2 years of screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11-06 (Actual); Primary Completion 2010-04-06 (Actual); Study Completion 2010-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=1064-003&kw=1064-003&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 4 treatment sequences of single doses of MK-1064 or placebo, administered over 4 study periods in a crossover design; then in Period 5 participants received, according to separate randomization, either a single dose of 20 mg MK-6096 or placebo, in an 18:2 ratio for overall study population.
Groups:
- MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4): Period 1 - single dose of 50 mg MK-1064, Period 2 - single dose of 250 mg MK-1064, Period 3 - single dose of placebo, Period 4 - single dose of 120 mg MK-1064.
- MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4): Period 1 - single dose of placebo, Period 2 - single dose of 50 mg MK-1064, Period 3 - single dose of 120 mg MK-1064, Period 4 - single dose of 250 mg MK-1064.
- MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4): Period 1 - single dose of 120 mg MK-1064, Period 2 - single dose of placebo, Period 3 - single dose of 250 mg MK-1064, Period 4 - single dose of 50 mg MK-1064.
- MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4): Period 1 - single dose of 250 mg MK-1064, Period 2 - single dose of 120 mg MK-1064, Period 3 - single dose of 50 mg MK-1064, Period 4 - single dose of placebo.
- MK-6096 20 mg (Period 5): Participants in this arm had completed the first 4 study periods, and were randomized to receive a single dose of 20 mg of MK-6096 in Period 5.
- Placebo (Period 5): Participants in this arm had completed the first 4 study periods, and were randomized to receive a single dose of placebo in Period 5.
Period: Period 1 - MK-1064 or Placebo
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After Period 1
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - MK-1064 or Placebo
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After Period 2
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - MK-1064 or Placebo
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After Period 3
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - MK-1064 or Placebo
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout After Period 4
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 5 | 5 | 5 | 5 | 0 | 0
Completed | 5 | 4 | 4 | 4 | 0 | 0
Not Completed | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0
Period: Period 5 - MK-6096 or Placebo
Arm/Group | MK-1064: 50 mg→250 mg→Placebo→120 mg (Period 1-4) | MK-1064: Placebo→50 mg→120 mg→250 mg (Period 1-4) | MK-1064: 120 mg→Placebo→250 mg→50 mg (Period 1-4) | MK-1064: 250 mg→120 mg→50 mg→Placebo (Period 1-4) | MK-6096 20 mg (Period 5) | Placebo (Period 5)
Started | 0 (In Period 5, participants previously in this arm appear in MK-6096 20 mg/Placebo (Period 5) arms) | 0 (In Period 5, participants previously in this arm appear in MK-6096 20 mg (Period 5) arm) | 0 (In Period 5, participants previously in this arm appear in MK-6096 20 mg (Period 5) arm) | 0 (In Period 5, participants previously in this arm appear in MK-6096 20 mg (Period 5) arm) | 16 (Participants entering Period 5 were previously in MK-1064/Placebo (Period 1-4) arms) | 1 (Participants entering Period 5 were previously in MK-1064/Placebo (Period 1-4) arms)
Completed | 0 | 0 | 0 | 0 | 14 (The 2 participants who did not complete Period 5 did not receive study drug in Period 5) | 1
Not Completed | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.60) [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Latency to Persistent Sleep (LPS) Following Single Doses of MK-1064 and Placebo
Description: LPS is measured during overnight sleep laboratory (polysomnography [PSG]) assessment and is defined as the duration of time from the beginning of PSG assessment to the first interval of 10 consecutive minutes of sleep.
Time Frame: 1 to 9 hours post dose, within each treatment period
Population: Per-Protocol. Note: Data included are those obtained from subjects during administration of MK-1064 doses in Period 1-4 and during administration of placebo in Period 1-4
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Groups:
- MK-1064 50 mg: Single dose of 50 mg MK-1064
- MK-1064 120 mg: Single dose of 120 mg MK-1064
- MK-1064 250 mg: Single dose of 250 mg MK-1064
- Placebo: Single dose of placebo
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 4.27 [2.34 to 7.78] | 3.68 [2.01 to 6.71] | 2.67 [1.46 to 4.88] | 17.93 [9.82 to 32.73]
Statistical Analysis 1: Comparison: MK-1064 50 mg vs Placebo; Analysis used a step-down approach. Mean log treatment difference of the highest MK-1064 dose versus placebo (MK-1064 - placebo) and 90% confidence interval (CI) were computed and back-transformed to obtain the 90% CI interval for LPS treatment ratio. If the CI lies completely below 1, testing continued to next lower MK-1064 dose. The hypothesis that MK-1064 is superior to placebo in decreasing LPS was supported if the CI lies below 1 for at least one dose; Test type: Superiority or Other; Geometric Mean Ratio = 0.24, 90% CI 2-sided [0.12 to 0.47] — Ratio is MK-1064/placebo
Statistical Analysis 2: Comparison: MK-1064 120 mg vs Placebo; Analysis used a step-down approach. Mean log treatment difference of the highest MK-1064 dose versus placebo (MK-1064 - placebo) and 90% CI were computed and back-transformed to obtain the 90% CI interval for LPS treatment ratio. If the CI lies completely below 1, testing continued to next lower MK-1064 dose. The hypothesis that MK-1064 is superior to placebo in decreasing LPS was supported if the CI lies below 1 for at least one dose; Test type: Superiority or Other; Geometric Mean Ratio = 0.21, 90% CI 2-sided [0.10 to 0.41] — Ratio is MK-1064/placebo
Statistical Analysis 3: Comparison: MK-1064 250 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric Mean Ratio = 0.15, 90% CI 2-sided [0.08 to 0.30] — Ratio is MK-1064/placebo

2. Primary Outcome: LPS Following Single Doses of MK-6096 and Placebo
Description: LPS is measured during overnight sleep laboratory (PSG) assessment and is defined as the duration of time from the beginning of PSG assessment to the first interval of 10 consecutive minutes of sleep.
Time Frame: 1 to 9 hours post dose, within each treatment period
Population: Per-Protocol. Note: Data included are those obtained from subjects during MK-6096 dose in Period 5 and during administration of placebo in any period. 1 subject took placebo within Periods 1-4 and also in Period 5. Data for both administrations of placebo are included (i.e., for placebo, analysis includes 21 observations from 20 subjects)
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Groups:
- MK-6096 20 mg: Single dose of 20 mg MK-6096
Arm/Group | MK-6096 20 mg | Placebo
Number analyzed (Participants) | 14 | 20
minutes | 0.87 [0.39 to 1.93] | 17.79 [9.21 to 34.35]
Statistical Analysis 1: Comparison: MK-6096 20 mg vs Placebo; Mean log treatment difference of MK-6096 versus placebo (MK-6096 - placebo) and 90% CI were computed and back-transformed to obtain the 90% CI interval for LPS treatment ratio; Test type: Superiority or Other; Geometric Mean Ratio = 0.05, 90% CI 2-sided [0.02 to 0.11] — Ratio is MK-6096/placebo

3. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study drug, is also an AE.
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 42 days)
Population: All Participants as Treated - all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | MK-6096 20 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 14 | 20
participants | 4 | 4 | 7 | 3 | 3

4. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 3
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 42 days)
Population: All Participants as Treated - all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | MK-6096 20 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 14 | 20
participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Wake Time After Sleep Onset (WASO) Following Single Doses of MK-1064 and Placebo
Description: WASO is measured during overnight sleep laboratory (PSG) assessment and is defined as the duration of wakefulness from the onset of persistent sleep (i.e., 10 consecutive minutes of sleep) to the end of PSG assessment the following morning.
Time Frame: 1 to 9 hours post dose, within each treatment period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
minutes | 22.41 [17.69 to 28.40] | 18.01 [14.21 to 22.82] | 19.90 [15.70 to 25.21] | 26.41 [20.84 to 33.46]
Statistical Analysis 1: Comparison: MK-1064 50 mg vs Placebo; Analysis used a step-down approach. Mean log treatment difference of the highest MK-1064 dose versus placebo (MK-1064 - placebo) and 90% CI were computed and back-transformed to obtain the 90% CI interval for WASO treatment ratio. If the CI lies completely below 1, testing continued to next lower MK-1064 dose. The hypothesis that MK-1064 is superior to placebo in decreasing WASO was supported if the CI lies below 1 for at least one dose; Test type: Superiority or Other; Geometric Mean Ratio = 0.85, 90% CI 2-sided [0.67 to 1.07] — Ratio is MK-1064/placebo
Statistical Analysis 2: Comparison: MK-1064 120 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 0.68, 90% CI 2-sided [0.54 to 0.86] — Ratio is MK-1064/placebo
Statistical Analysis 3: Comparison: MK-1064 250 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 0.75, 90% CI 2-sided [0.60 to 0.95] — Ratio is MK-1064/placebo

6. Secondary Outcome: WASO Following Single Doses of MK-6096 and Placebo
Description: as for outcome 5
Time Frame: 1 to 9 hours post dose, within each treatment period
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | MK-6096 20 mg | Placebo
Number analyzed (Participants) | 14 | 20
minutes | 16.65 [12.91 to 21.48] | 26.41 [21.17 to 32.95]
Statistical Analysis 1: Comparison: MK-6096 20 mg vs Placebo; Mean log treatment difference of MK-6096 versus placebo (MK-6096 - placebo) and 90% CI were computed and back-transformed to obtain the 90% CI interval for WASO treatment ratio; Test type: Superiority or Other; Geometric Mean Ratio = 0.63, 90% CI 2-sided [0.50 to 0.79] — Ratio is MK-6096/placebo

7. Secondary Outcome: Change From Baseline in Choice Reaction Time (CRT) Following Single Doses of MK-1064 and Placebo
Description: CRT assessment used in this study is a two-choice, computer-controlled test in which the participant responds to stimulus words presented on the screen of a laptop computer. During the test either the word "NO" or the word "YES" is presented on the screen and the participant is instructed to press the corresponding button as quickly as possible. There are 50 trials for which each stimulus word is chosen randomly with equal probability and there is a varying inter-stimulus interval. The mean reaction time of accurate responses is determined. The assessment is performed pre-dose and at 10 hours post dose. The outcome measure is change from baseline to post dose in reaction time.
Time Frame: Pre-dose and 10 hours post dose, within each treatment period
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
milliseconds
  Baseline (Pre-dose) | 408.79 [390.94 to 426.64] | 423.39 [400.05 to 446.72] | 418.83 [399.44 to 438.22] | 414.85 [392.90 to 436.79]
  Change at 10 hours post dose | 17.25 [4.41 to 30.10] | 19.94 [7.10 to 32.78] | 21.04 [8.20 to 33.88] | 14.66 [1.82 to 27.50]
Statistical Analysis 1: Comparison: MK-1064 50 mg vs Placebo; Analysis used a step-up approach. Mean treatment difference in change from baseline of the lowest MK-1064 dose versus placebo (MK-1064 - placebo) and 90% CI were computed. If the CI lies completely below 25 milliseconds, testing continued to the next higher MK-1064 dose. The hypothesis that at least one dose of MK-1064 does not produce psychomotor impairment versus placebo as assessed by CRT will be supported if the CI lies below 25 milliseconds for at least one dose; Test type: Superiority or Other; Mean Difference (Final Values) = 2.59, 90% CI 2-sided [-12.01 to 17.20] — Difference is MK-1064 - placebo
Statistical Analysis 2: Comparison: MK-1064 120 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.28, 90% CI 2-sided [-9.33 to 19.88] — Difference is MK-1064 - placebo
Statistical Analysis 3: Comparison: MK-1064 250 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.38, 90% CI 2-sided [-8.23 to 20.98] — Difference is MK-1064 - placebo

8. Secondary Outcome: Change From Baseline in CRT Following Single Doses of MK-6096 and Placebo
Description: as for outcome 7
Time Frame: Pre-dose and 10 hours post dose, within each treatment period
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | MK-6096 20 mg | Placebo
Number analyzed (Participants) | 14 | 20
milliseconds
  Baseline (Pre-dose) | 425.94 [391.76 to 460.12] | 417.81 [396.11 to 439.51]
  Change at 10 hours post dose | 24.04 [8.04 to 40.04] | 14.74 [1.49 to 27.99]
Statistical Analysis 1: Comparison: MK-6096 20 mg vs Placebo; Mean treatment difference in change from baseline of MK-6096 versus placebo (MK-6096 - placebo) and 90% CI were computed; Test type: Superiority or Other; Mean Difference (Final Values) = 9.30, 90% CI 2-sided [-7.10 to 25.70] — Difference is MK-6096 - placebo

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (Up to approximately 42 days)
Description: Analysis population is All Participants as Treated, defined as all participants who received at least one dose of study drug
Arm/Group | MK-1064 50 mg | MK-1064 120 mg | MK-1064 250 mg | MK-6096 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 2/20 | 5/20 | 3/14 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1064 50 mg (N=20) | MK-1064 120 mg (N=20) | MK-1064 250 mg (N=20) | MK-6096 20 mg (N=14) | Placebo (N=20)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.